CLINICAL TRIAL: NCT03757780
Title: Association of Low Birth Weight Fetuses With Caffeine Use
Brief Title: Low Birth Weight Fetuses With Caffeine Use
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: low birth weight
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Low; Birthweight, Extremely (999 Grams or Less)
MeSH Terms: conditions — Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant ladies who are caffeine using: ladies who uses caffeine during pregnancy
  Interventions: Other: Questionaire

INTERVENTIONS:
Other: Questionaire — A questionaire will be made to pregnant ladies who take caffeine during pregnancy

SUMMARY:
Globally, it has been estimated that 15.5% of all infantsare born low birth weight, defined as birthweight less than 2,500 g .

DETAILED DESCRIPTION:
Low birth weight is not only associated with neonatal mortality and morbidity.

but also with a higher risk of chronic diseases such as type 2 diabetes and cardiovascular diseases in adult life

ELIGIBILITY:
Inclusion Criteria:

* Age group: 18-40
* Pregnant females attending regular post-natal care visits

Exclusion Criteria:

* • Female patients with other acute or chronic illness

  * Cardiovascular disease
  * Neoplasms
  * Current diabetes mellitus, pregnancy induced diabetes
  * Renal impairment (serum creatinine 120 mol/liter), and hypertension (blood pressure 140/85 mm Hg).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — • pregnant women with age group between : 18-40
Study Population: Age group: 18-40
  •Pregnant females attending regular post-natal care visits
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-15 (Estimated)

PRIMARY OUTCOMES:
The number of pregnant ladies who will have low birth weight babies | within 2 months
  Mothers who will give birth to low birth weight infants

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Study Chair — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah and Kasralainy hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No